CLINICAL TRIAL: NCT05309343
Title: Cohort Study on Treatment of Cardiovascular Diseases With Traditional Chinese Medicine
Acronym: CSCD-TCM plus
Status: Recruiting | Type: Observational
Sponsor: Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Lin Li, researcher, Tianjin University of Traditional Chinese Medicine
Other Study IDs: CSCD-TCM plus
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, feces, saliva, tongue coating
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Western medicine treatment with Chinese medicine treatmen
  Interventions: Drug: Chinese patent medicine
- Non-exposed group: Western medicine treatment

INTERVENTIONS:
Drug: Chinese patent medicine — Shexiang Baoxin Pill, Tongxinluo Capsule, Tongmai Yangxin Pill, Xuefu Zhuyu Capsule, Qishen Yiqi Dropping Pill, etc.
  Groups: Exposed group

SUMMARY:
This is a cohort study performed in patients with cardiovascular diaeases who were treated with oral Chinese medicine and Western medicine. Collect indicators such as the incidence of cardiovascular events, all due to readmission, all due to death. To hospital using clinical samples to detect genomics, proteomics, metabolomics, intestinal flora and sclerotia.To explore the clinical efficacy of Chinese patent medicine in the treatment of cardiovascular diseases, and provide reliable data support for its clinical application.

ELIGIBILITY:
Inclusion Criteria:

All patients admitted to the Department of Cardiovascular Medicine at The First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, The Second Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin Chest Hospital, Tianjin Hospital of ITCWM Nankai Hospital and Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital were considered for inclusion in this study, and all Western medical diagnoses were identified and classified according to the International Classification of Diseases, 11th Revision (ICD-11).

Exclusion Criteria:

No exclusion criteria.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The collaboration network of coronary heart disease research medical units formed by the research group, including The First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, The Second Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin Chest Hospital, Tianjin Hospital of ITCWM Nankai Hospital and Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital#a total of 6 hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Events Cardiovascular Events Cardiovascular Events | one year
  Non-fatal myocardial infarction, non-fatal ischemic stroke, unplanned hemodynamic reconstruction.
All due to readmission | one year
  Readmission for cardiovascular events and readmission for other reasons.
All due to death | one year
  Cardiac death and death from other causes.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin University of Traditional Chinese Medicine, Tianjin, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Yang T, Zheng H, Pan G, Guo R, Liu F, Liu S, Tao S, Li L, Yang R, Yu C. Relationship between the circulating N-terminal pro B-type natriuretic peptide and the risk of carotid artery plaque in different glucose metabolic states in patients with coronary heart disease: a CSCD-TCM plus study in China. Cardiovasc Diabetol. 2023 Nov 2;22(1):299. doi: 10.1186/s12933-023-02015-y. PMID 37919791